CLINICAL TRIAL: NCT03670056
Title: A Pilot Study of Combination Immunotherapy With Ipilimumab and Nivolumab in Patients With Recurrent Extensive Stage Small Cell Lung Cancer (SCLC) Who Have Previously Received Platinum-based Chemotherapy
Brief Title: Ipilimumab and Nivolumab in Recurrent Extensive Stage Small Cell Lung Cancer After Receiving Platinum-based Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Anne Chiang, Principal Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023361; CA209-9YT (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer
Keywords: combination immunotherapy; platinum-based chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Patients will be treated with nivolumab 1 mg/kg and ipilimumab 3 mg/kg, starting on Day 1. Patients will receive 4 doses of each nivolumab and ipilimumab and then will receive nivolumab 240 mg starting week 13 (day 85) every 2 weeks until progression, unacceptable toxicity, withdrawal of consent, or the study ends, whichever occurs first.
  Interventions: Drug: Combination immunotherapy with Ipilimumab and Nivolumab

INTERVENTIONS:
Drug: Combination immunotherapy with Ipilimumab and Nivolumab — Patients will be treated with nivolumab 1 mg/kg and ipilimumab 3 mg/kg, starting on Day 1. Patients will receive 4 doses of each nivolumab and ipilimumab and then will receive nivolumab 240 mg starting week 13 (day 85) every 2 weeks until progression, unacceptable toxicity, withdrawal of consent, or the study ends, whichever occurs first.

SUMMARY:
This is a pilot study of patients who previously received platinum chemotherapy with recurrent SCLC to evaluate the change in the ratio of intratumoral Teff/Treg cells and clinical benefit of treatment with nivolumab and ipilimumab.

DETAILED DESCRIPTION:
The primary objective of this study is t assess whether the change in the ratio of effector T cells (Teff) to regulatory T cells (Treg), i.e. CD8 positive/FoxP3 expressing CD4 T cells, between pre- and on- treatment biopsies, will predict clinical response in patients with recurrent SCLC treated with combination therapy with nivolumab and ipilimumab.

Secondary objectives of the study include: to determine the objective response rate per RECIST 1.1 and immune-related response criteria, duration of response, progression free survival, and overall survival with nivolumab and ipilimumab in patients with recurrent SCLC; to evaluate changes in the tumor immune microenvironment and blood after treatment with ipilimumab and nivolumab; and to evaluate circulating tumor DNA (ctDNA) as a marker for response to therapy.

ELIGIBILITY:
Inclusion:

* Patients with an active autoimmune disease requiring systemic treatment within the past 3 months, or a syndrome that requires systemic steroids greater than dexamethasone 2 mg daily (or equivalent) or immunosuppressive agents within the past 3 months will be ineligible. Patients with a documented history of severe autoimmune disease but have been off of steroids and immunosuppressive agents for greater than 3 months, or only require intermittent steroid bursts may be eligible following discussion and approval from the Principal Investigator. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects who require intermittent use of inhaled steroids or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement, or psoriasis not requiring systemic therapy (within the past 3 years) or Type 1 diabetes on stable insulin will not be excluded from the study
* Histologically or cytologically documented Extensive Stage Small Cell Lung Cancer with documented disease progression after at least one prior systemic regimen, including one platinum-based regimen, with progression of disease on or after their most recent therapy. Patients previously diagnosed with limited stage Small Cell Lung Cancer treated with concurrent chemoradiation with a platinum doublet now diagnosed with recurrent extensive disease are eligible.
* ECOG performance status of 0 to 2
* Measurable disease with at least one tumor site amenable to biopsy
* Patients may have untreated asymptomatic Central Nervous System (CNS) metastases or treated CNS metastases if they are not currently receiving corticosteroids greater than dexamethasone 2 mg daily or equivalent for 7 days prior to the first dose of study drug. Patients should have completed stereotactic radiation or whole-brain radiation at least 2 weeks prior to Cycle 1, Day 1

Exclusion:

* Patients with an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids > dexamethasone 2 mg daily (or equivalent dose of other corticosteroids) or other immunosuppressive agents.
* Treatment with systemic immunosuppressive medications including but not limited to, dexamethasone at doses > 2 mg or equivalent dose of other corticosteroids, cyclophosphamide, tacrolimus, sirolimus, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor (anti-TNF) agents within 2 weeks prior to initiation of trial therapy. Inhaled or topically applied steroids, and acute and chronic standard-dose NSAIDs are permitted. Replacement steroids are also permitted.
* Prior treatment with anti-CTLA4 antibodies. Prior anti-PD1 or anti-PDL1 therapy is allowed.
* Symptomatic untreated CNS metastases. Patients with asymptomatic CNS metastases are eligible. Patients with symptomatic brain metastases are eligible, provided they meet all of the following criteria:

  * Completed stereotactic radiosurgery or whole- brain radiation at least 2 weeks prior to Cycle 1, Day 1.
  * No evidence of interim progression between the completion of CNS-directed therapy and the start of trial therapy.
  * No ongoing requirement for steroids greater than dexamethasone 2 mg daily (or equivalent dose of other corticosteroids) as therapy for CNS disease; anticonvulsants at a stable dose are allowed.
* History of leptomeningeal carcinomatosis.
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Any systemic anti-cancer chemotherapy, within 21 days prior to initiation of study treatment.
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 21 days prior to enrollment.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery or traumatic injury within 4 weeks of starting study drug.
* - Women who are pregnant or lactating.
* - Known infection with HIV, HBV or HCV. Patients with prior exposure to hepatitis, but no evidence of active or chronic infection, may be eligible.
* - Evidence of end-organ damage as defined by the following laboratory results obtained within 14 days prior to the first study treatment:

  * ANC <1,000 cells/µL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1).
  * Platelet count <75,000/µL (without transfusion within 2 weeks prior to Cycle 1, Day 1).
  * Hemoglobin <8.0 g/dL (Patients may be transfused to meet this criterion).
  * AST and ALT ≥2.5 x ULN, with the following exceptions: Patients with documented liver metastases: AST and/or ALT≥5 x ULN. o Serum bilirubin ≥1.5 x ULN (Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled).
  * INR and aPTT ≥1.5 x ULN (This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the ratio of Teff/Treg cells | Up to 24 months
  The primary analysis will use the nonparametric Mann-Whitney sign test to compare the change in the ratio of Teff/Treg cells in those patients who respond or not to treatment. This test compares the rate of response in those with above and below Teff/Treg ratio.

SECONDARY OUTCOMES:
Response rate | Up to 24 months
  Objective response is defined as a complete or partial response, as determined by investigator assessment using RECIST v1.1 and immune-related response criteria (irRC) . Response will be confirmed by repeat assessments ≥4 weeks after initial documentation. Patients not meeting these criteria, including patients without any post baseline tumor assessment, will be considered non-responders in the analysis of objective response.
Duration of response | Up to 24 months
  Duration of response is defined as the time from the initial complete or partial response to the time of disease progression or death, whichever occurs first. If a patient does not experience death or disease progression before the end of the study, duration of response will be censored at the day of the last tumor assessment. If no tumor assessments were performed after the date of the first occurrence of a complete or partial response, duration of objective response will be censored at the date of the first occurrence of a complete or partial response plus 1 day.
Progression-free survival | Up to 24 months
  Progression-free survival (PFS) is defined as the time from the first day of treatment until progression of disease using RECIST v1.1 and immune-related response criteria (irRC) . If a patient has not experienced progressive disease or death, PFS will be censored at the day of the last tumor assessment. Patients with no post baseline tumor assessments will be censored at the date of first study treatment plus 1 day.

OTHER OUTCOMES:
Change in ctDNA | Up to 24 months
  Circulating tumor DNA (ctDNA) will be collected throughout the trial, including at 4 weeks, at the time of repeat biopsy. We will assess if the change in variant allele frequencies from baseline sample to the 4 week sample predicts response to therapy and correlate to objective response rate.
Change in tumor microenvironment | Up to 24 months
  Immunohistochemistry (IHC) and quantitative measurement (QiF) of fluorescent signals of tumor infiltrating lymphocytes after immunofluorescence staining of pre- and on-treatment biopsy samples will be used. The baseline and change in tumor microenvironment using IHC and QIF for tumor infiltrating lymphocytes will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chiang, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No